CLINICAL TRIAL: NCT04378543
Title: A Phase 1b/2a Safety Evaluation of ART352-L in Subjects Undergoing Posterolateral Spinal Fusion
Brief Title: Safety Evaluation of ART352-L in Subjects Undergoing Posterolateral Spinal Fusion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankasa Regenerative Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART-SPF-ART352L-001
Record Dates: First submitted 2020-04-30; First posted 2020-05-07 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Degenerative Spondylolisthesis
Keywords: spine; spondylolisthesis; degenerative disc disease; back pain
MeSH Terms: conditions — Spondylolisthesis; Intervertebral Disc Degeneration; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ART252-L (Experimental): local autologous bone graft will be treated ex vivo once with ART352-L prior to re-implantation into the site of spinal fusion
  Interventions: Biological: ART352-L

INTERVENTIONS:
Biological: ART352-L — recombinant human Wnt3a protein delivered on liposomes to local autologous bone graft during posterolateral fusion procedures

SUMMARY:
Ankasa Regenerative Therapeutics, Inc. (Ankasa) is developing ART352-L, a liposomal formulation of recombinant human Wnt3A protein, that is applied ex vivo, to harvested autologous bone grafts (autograft) to enhance the osteogenic properties of the autograft prior to reimplantation in orthopedic surgeries.

This is a phase 1/2 open label safety evaluation of ART352-L treated autologous bone grafts in patients undergoing posterolateral lumbar spinal fusion to treat single level degenerative spondylolisthesis. The primary objective of the study is to evaluate the safety and tolerability of ART352-L treated local bone autografts in patients being treated for this condition, with the secondary objective to evaluate the rates of early and overall spinal fusion. Additionally, changes in patient mobility and quality of life measures from baseline following treatment with ART352-L will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥50 years of age scheduled to undergo single level posterolateral lumbar spinal fusion surgery in conjunction with local autograft bone for degenerative spondylolisthesis
2. Psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent
3. Willing and able to undergo diagnostic imaging, inclusive of X-rays and CT scans with contrast
4. Persistent, disabling pain after at least 6 months of non-surgical intervention (e.g., anti-inflammatory medication, physical therapy, chiropractic care) prior to providing informed consent
5. Pre-operative Oswestry Disability Index (ODI) Score ≥30
6. Grade 1 or less spondylolisthesis or retrolisthesis
7. Absence of neurological motor deficit
8. Agree to use a highly reliable method of birth control (male and female subjects) for at least 90 days after administration of Investigational Product (IP) - Women of childbearing potential must have a negative pregnancy test at screening and again ≤7 days prior to surgery. Perimenopausal women must be amenorrheic for at least 12 months prior to the time of providing informed consent to be considered of non-childbearing potential.
9. Agree to remain nicotine-free for the duration of their participation in the study

Exclusion Criteria:

1. Multiple level spondylolistheses or a primary diagnosis of low back pain syndrome secondary to diseases other than degenerative spondylolisthesis
2. Concurrent medications that affect bone homeostasis including, but not limited to, bisphosphonates
3. Ongoing / existing infections in or around the surgical site or spine
4. Prior lumbar spine arthrodesis
5. Concurrent clinically significant autoimmune disorder or systemic inflammatory disease
6. Known hypersensitivity to recombinant Wnt proteins
7. Use of tobacco; subjects must be nicotine-free at screening and agree to remain nicotine free for the duration of the study
8. Use of medications that may impair cell proliferation and bone healing including: chemotherapy, radiation, chronic steroids and immunosuppressive drugs. Note: Medications that may impair cell proliferation are to be discussed with the protocol medical monitor prior to enrollment
9. Severe established osteoporosis requiring active treatment e.g., with bone density more than 2.5 standard deviations below the young adult mean with one or more osteoporotic fractures
10. A Body Mass index (BMI) ≥ 40 unless documentation clearly demonstrates why BMI is not a primary factor in the subject's decreased mobility
11. Chronic opioid use
12. History of deep vein thrombosis (DVT) or blood clotting abnormalities
13. Uncontrolled diabetes mellitus
14. Pre-operative/anesthesia evaluations deeming the subject ineligible for surgery
15. Female subjects who are pregnant or intend to become pregnant during the course of the study
16. Male subjects, if not infertile or surgically sterilized, who will not agree to use highly-effective contraception or to not donate sperm from screening until at least 90 days after receiving IP
17. Active malignancy ≤5 years prior to providing informed consent. EXCEPTIONS: Non-melanotic skin cancer, carcinoma-in-situ of the cervix. NOTE: If there is a history of prior malignancy, the subject must not be receiving other specific treatment for their cancer.
18. Concurrent participation in another investigational drug, biologic or device study that could confound study data
19. Involvement in or plans to engage in litigation or receiving Worker's Compensation related to neck, back, or leg pain

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 weeks
  Incidence of adverse events and adverse events of special interest
Safety and Tolerability | 8 weeks
  Incidence of adverse events and adverse events of special interest
Safety and Tolerability | 26 weeks
  Incidence of adverse events and adverse events of special interest
Safety and Tolerability | 52 weeks
  Incidence of adverse events and adverse events of special interest
Safety and Tolerability | 104 weeks
  Incidence of adverse events and adverse events of special interest

SECONDARY OUTCOMES:
Rate of early fusion | 26 weeks
  Rate of early fusion using Lenke scoring of computed tomography (CT) scans
Rate of fusion | 52 weeks
  Rate of fusion using Lenke scoring of CT scans
Rate of fusion | 104 weeks
  Rate of fusion using Lenke scoring of CT scans
Oswestry Disability Index | 8 weeks
  Change from baseline in Oswestry Disability Index
Oswestry Disability Index | 26 weeks
  Change from baseline in Oswestry Disability Index
Oswestry Disability Index | 52 weeks
  Change from baseline in Oswestry Disability Index
Oswestry Disability Index | 104 weeks
  Change from baseline in Oswestry Disability Index
Short Form-36 (SF-36) | 8 weeks
  Change from baseline in Short Form-36 (SF-36) score
Short Form-36 (SF-36) | 26 weeks
  Change from baseline in Short Form-36 (SF-36) score
Short Form-36 (SF-36) | 52 weeks
  Change from baseline in Short Form-36 (SF-36) score
Short Form-36 (SF-36) | 104 weeks
  Change from baseline in Short Form-36 (SF-36) score
Visual Analog Scale (VAS) Pain | 8 weeks
  Change from baseline in Visual Analog Scale (VAS) Pain assessment
Visual Analog Scale (VAS) Pain | 26 weeks
  Change from baseline in Visual Analog Scale (VAS) Pain assessment
Visual Analog Scale (VAS) Pain | 52 weeks
  Change from baseline in Visual Analog Scale (VAS) Pain assessment
Visual Analog Scale (VAS) Pain | 104 weeks
  Change from baseline in Visual Analog Scale (VAS) Pain assessment
Patient Reported Outcomes Measurement Information System (PROMIS) - Global 10 | 8 weeks
  Change from baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Global-10 Score
Patient Reported Outcomes Measurement Information System (PROMIS) - Global 10 | 26 weeks
  Change from baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Global-10 Score
Patient Reported Outcomes Measurement Information System (PROMIS) - Global 10 | 52 weeks
  Change from baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Global-10 Score
Patient Reported Outcomes Measurement Information System (PROMIS) - Global 10 | 104 weeks
  Change from baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Global-10 Score

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Keck School of Medicine, University of Southern California, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - Wexner Medical Center, The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No